CLINICAL TRIAL: NCT02087189
Title: TD01 Master Study (Safety and Efficacy Study)
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: TA107
Record Dates: First submitted 2014-03-04; First posted 2014-03-14 (Estimated); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2020-01

CONDITIONS: ICD/CRT-D Indication
Keywords: ICD, CRT-D, lead

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD/ CRT-D therapy
  Interventions: Device: First ICD/CRT-D implantation or upgrade from pacemaker

INTERVENTIONS:
Device: First ICD/CRT-D implantation or upgrade from pacemaker
  Other Names: TD01 (investigational device); Lumax 540, 640 or 740: VR-T, DR-T or HF-T or; Ilesto 5 or Ilesto 7 DF-1: VR-T, DR-T or HF-T or; Iforia 3, 5 or Iforia 7 DF-1: VR-T, DR-T or HF-T; (or successor); Free choice of additional RA and/or LV lead (if applicable)

SUMMARY:
This clinical investigation is designed to confirm the safety and efficacy of the TD01 ICD lead.

ELIGIBILITY:
Inclusion Criteria:

* Meet standard indication for ICD/CRT-D therapy
* First ICD/CRT-D implantation or upgrade from pacemaker
* Duly signed informed consent form
* Willing to participate for the whole study duration
* Patient accepts Home Monitoring concept and is able to activate and use the CardioMessenger
* Patient has a legal capacity and ability to consent

Exclusion Criteria:

* Meet a standard contraindication for an ICD/CRT-D therapy
* Age < 18 years
* Pregnant or breast-feeding
* Cardiac surgery planned within the next six months
* Enrollment in another cardiac clinical investigation with active treatment arm
* Mechanical tricuspid valve prosthesis or severe tricuspid valve disease
* Known dexamethasone acetate intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected for the investigation should be from the investigator's general patient population according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Gunkel, Dr. med., Principal Investigator — Coordinating Investigator, former PI at the Klinikum Frankfurt (Oder)
Locations (5):
- Kepler Universitätsklinikum, Linz, Austria
- Germany (4):
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder), Brandenburg
  - Vivantes-Krankenhaus Neukölln, Berlin
  - DRK Krankenhaus Chemnitz-Rabenstein, Chemnitz
  - Kliniken im Naturpark Altmühltal, Kösching

RESULTS

PARTICIPANT FLOW:
Groups:
- ICD/ CRT-D Therapy With TD01 as ICD Lead: enrolled as a patient planned with ICD and TD01 implantation
Period: Overall Study
Arm/Group | ICD/ CRT-D Therapy With TD01 as ICD Lead
Started | 30
Completed | 28
Not Completed | 2
Not completed — enrolled but did not receive a TD01 as implant | 2

BASELINE CHARACTERISTICS:
Population: analysis include only the 28 patients that received the TD01 as implant
Groups:
- ICD/ CRT-D Therapy With TD01 as ICD Lead: patients with TD01 as implanted ICD lead
Arm/Group | ICD/ CRT-D Therapy With TD01 as ICD Lead
Number analyzed (Participants) | 28
Age, Continuous [Median (Standard Deviation); unit: years] | 70.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 21
Weight [Median (Standard Deviation); unit: kg] | 84.5 (19.8)
Height [Median (Standard Deviation); unit: cm] | 172.0 (8.2)
Body Mass Index (BMI) [Median (Standard Deviation); unit: kg/m²] | 28.5 (5.1)
Left Ventricular Ejection Fraction (LVEF) [Median (Standard Deviation); unit: %] — LVEF is calculated by dividing the volume of blood pumped from the left ventricle per beat (stroke volume) by the volume of blood collected in the left ventricle at the end of diastolic filling (end-diastolic volume).
  % | 30 (12.7)
NYHA class [Number; unit: participants] — Class I: Ordinary physical activity does not cause undue dyspnea or fatigue. Class II: Comfortable at rest. Ordinary physical activity results in dyspnea or fatigue.
  Class III: Comfortable at rest. Less than ordinary physical activity results in dyspnea or fatigue.
  Class IV: Symptoms of heart failure may be present even at rest. If any physical activity is undertaken, discomfort is increased.
  participants
    NYHA class I | 2
    NYHA class II | 11
    NYHA class III | 15
    NYHA class IV | 0

OUTCOME MEASURES:

1. Primary Outcome: TD01 Pacing Threshold
Description: Non-inferiority of the pacing threshold compared to Linox TD. It is expected, that pacing thresholds of the TD01 leads will be statistically significant lower than 0.8V.
  Pacing threshold is the minimal electrical stimulus (voltage) required to produce consistent cardiac depolarization (heart contraction). Linox TD is another (predecessor) electrode that is used for comparison.
Time Frame: 3 month follow-up
Population: per protocol analysis
Measure: Median (95% Confidence Interval); unit: V
Arm/Group | ICD/ CRT-D Therapy With TD01 as ICD Lead
Number analyzed (Participants) | 20
V | 0.5 [0.3 to 0.6]

2. Primary Outcome: TD01 Sensing Amplitude
Description: Non-inferiority of the sensing amplitude compared to Linox TD. It is expected, that the sensing amplitudes of the TD01 leads will be statistically significant higher than 9.7mV.
  Sensing amplitude is the value for the measured voltage maximum (mV) during the ventricular depolarization (QRS complex during contraction). Linox TD is another (predecessor) electrode that is used for comparison.
Time Frame: 3 month follow-up
Population: per protocol analysis
Measure: Median (95% Confidence Interval); unit: mV
Arm/Group | ICD/ CRT-D Therapy With TD01 as ICD Lead
Number analyzed (Participants) | 20
mV | 19.6 [16.1 to 21.4]

3. Secondary Outcome: SADE-free Rate Related to TD01
Description: SADE-free rate related to TD01. It is expected, that the SADE-free rate is higher than 0.9 (90%).
  SADE Free Rate is a safety parameter and defined as p = 1 - number of SADEs divided by the number of TD01 leads implanted. Whereby Serious Adverse Device Effects (SADEs) are accounted that relate to the TD01 ICD lead and were observed between implantation until the predefined follow-up time, e.g. the three month follow-up.
Time Frame: 3 month follow-up
Population: full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ICD/ CRT-D Therapy With TD01 as ICD Lead
Number analyzed (Participants) | 28
percentage of participants | 96.4 [84.2 to 100]

ADVERSE EVENTS:
Time Frame: All AEs were systematically recorded for the first two years of patient follow-up. From 24-month follow-up until 60-month follow-up only SADEs related to the investigational device were required to be reported per protocol, but AE reporting remained possible.
Description: AE and SAE were defined according to ISO 14155:2011 in the study protocol.
Groups:
- ICD/ CRT-D Therapy With TD01 as ICD Lead: patient with TD01 as implanted ICD lead
Arm/Group | ICD/ CRT-D Therapy With TD01 as ICD Lead
All-Cause Mortality (participants affected / at risk) | 6/28
Serious Adverse Events (participants affected / at risk) | 19/28
Other Adverse Events (participants affected / at risk) | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICD/ CRT-D Therapy With TD01 as ICD Lead (N=28)
Adverse drug reaction (General disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 12 (12)
Cardiac failure chronic (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2)
Cataract (Eye disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic sinusitis (Infections and infestations) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Device lead damage (Product Issues) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Duodenal polyp (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Implant site haematoma (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Lead dislodgement (Product Issues) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Phlebitis (Vascular disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 3 (3)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 5 (5)
Rhinitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No